CLINICAL TRIAL: NCT00457535
Title: Recombinant Human Erythropoietin Dose, Serum Adiponectin, and All-Cause Mortality in Patients Beginning Hemodialysis
Brief Title: Study of the Relationship Between rHuEPO Dose, Serum ADPN, and Mortality in Patients Beginning HD
Status: Terminated | Type: Observational
Sponsor: Hamamatsu University (Other)
Collaborators: Shitoro Clinic (Unknown); Fujinomiya City Hospital (Other); Iwata City Hospital (Other); Seirei Mikatabara General Hospital (Unknown); Seirei Hamamatsu General Hospital (Other); Hamana Clinic (Other); Tadokoro Clinic (Unknown); Makoto Clinic (Unknown); Maruyama Memorial General Hospital (Other); Sun-Sanaru Clinic (Unknown)
Other Study IDs: 710808
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-04

CONDITIONS: Renal Dialysis
Keywords: recombinant human erythropoietin; adiponectin; mortality

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Responsiveness of recombinant human erythropoietin (rHuEPO) is known to be related with body fatness in hemodialysis (HD) patients. Adiponectin (ADPN) is inversely associated with body fat mass, and in healthy subjects, low ADPN is a predictor of mortality. Recently, higher rHuEPO dose itself is demonstrated to be associated with poor prognosis. So, in this study, we prospectively examined the relationship between rHuEPO dose, serum ADPN, and mortality in patients beginning HD.

DETAILED DESCRIPTION:
We selected 85 patients (51 men/34 women, age; 64±15 years) who survived for more than 3 months after the start of HD. After determining initial rHuEPO dosage, we followed the patients for 3 years, and examined an association between rHuEPO dose, serum ADPN, and all-cause mortality.

We could follow totally 74 out of 85 patients for 3 years; 59 patients were survived, but 15 patients expired. Dosage of rHuEPO was significantly and negatively correlated with body mass index (BMI) (r=-0.44, p<0.01) and positively with serum ADPN (r=0.29, p<0.02), but not with leptin. Cox-hazards regression analysis adjusted by age, sex and underlying kidney disease revealed that rHuEPO dose and serum ADPN, as well as nutritional parameter such as protein catabolic rate became significant determinants of 3-year mortality. There was a 12.7% risk increase for 10U/kg/week increase in rHuEPO dose and 1.3% increase for 1µg/ml increment of serum ADPN for the 3-year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients who had first started hemodialysis therapy from August 2000 to May 2001 in 11 dialysis centers in Shizuoka prefecture area.

Exclusion Criteria:

* nothing particular

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-08; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Naro Ohashi, MD,PhD, Principal Investigator — First Department of Medicine, Hamamatsu University School of Medicine